CLINICAL TRIAL: NCT03664973
Title: Effect of the Serratus Plane Block on the Outcome in Patient With Multiple Rib Fractures: A Prospective, Randomized, Controlled Trial
Brief Title: Serratus Plane Block for Rib Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Serratus GC
Record Dates: First submitted 2018-09-02; First posted 2018-09-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2019-05

CONDITIONS: Chest Trauma; Chest Pain
MeSH Terms: conditions — Thoracic Injuries; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous (Experimental): continuous local anesthetic infusion (ropivacaine 0.2%)on the serratus plane for at least 72h adds to a Single-shot serratus plane block with ropivacaine 0.37% solution 20 ml.
  Interventions: Procedure: Serratus plane block
- single-shot (Active Comparator): Single-shot serratus plane block with ropivacaine 0.37% solution 20 ml
  Interventions: Procedure: Serratus plane block

INTERVENTIONS:
Procedure: Serratus plane block — Local anesthetic infusion though a peripheral nerve catheter placed on the 5th rib under the serratus plane

SUMMARY:
Patients with ipsilateral multiple rib fractures will be randomized to receive either a single-shot ultrasound-guided serratus plane block, or a continuous serratus plane block within 24h from the chest trauma. Primary outcome is the difference in forced respiratory volume (FEV1) at 72h.

DETAILED DESCRIPTION:
Patients admitted in emergency department with a chest trauma and ipsilateral multiple rib fractures, will be randomized as described above. All patients will receive the serratus block with a ropivacaine 0.37% solution 20 ml. Then, they will randomized to receive either a peripheral catheter placed above the 5th rib on the middle axillary line, or nothing. In all patients postoperative analgesia also include Paracetamol 1g IV each 6h and a patient controlled analgesia (PCA) of morphine set out as follow: bolus 1 mg, loch out 15 min, max 4 boluses each hour. In all patients an arterial blood sample for gas analysis and a FEV1 will be achieved before the block, after 1 hour and at 72h.

ELIGIBILITY:
Inclusion Criteria:

* 2 o more ipsilateral rib fractures
* Trauma within 24h from hospital admission
* Informed consent

Exclusion Criteria:

* Chest drain
* head trauma
* bilateral rib fractures
* Intensive care admission

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary change function | day 0 and day 3
  FEV 1

SECONDARY OUTCOMES:
Numerical rating scale (NRS) of pain | day 0, day 1, day 2, day 3, day 4
  Pain both at rest and on movement on a 0-10 scale where 0 is the best and 10 the worst
Morphine | day 0, day 1, day 2, day 3, day 4
  morphine requirement
hospital stay | day 1, day 2, day 3, day 4, day 5, day 6, day7
  time to fill the discharge criteria

CONTACTS AND LOCATIONS:
Locations (1):
- AUSL IRCCS Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: Undecided